CLINICAL TRIAL: NCT03619174
Title: LIBERATE International: Evaluation of the Safety and Efficacy of the Viveve Treatment for Stress Urinary Incontinence
Brief Title: LIBERATE International
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Viveve Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIBERATE International
Record Dates: First submitted 2018-07-26; First posted 2018-08-07 (Actual); Results first posted 2022-08-18 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2019-07

CONDITIONS: Stress Urinary Incontinence
Keywords: incontinence; urine; urinary; pee; leak; SUI
MeSH Terms: conditions — Urinary Incontinence, Stress; Toxemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active Treatment (Active Comparator): Treatment dose
  Interventions: Device: Viveve Treatment
- Sham Treatment (Placebo Comparator): Sub-therapeutic dose
  Interventions: Device: Viveve Treatment

INTERVENTIONS:
Device: Viveve Treatment — The Viveve system is a monopolar radiofrequency system that uses surface cooling and radiofrequency (RF) energy delivery to provide a non-surgical and minimally-invasive approach to generate heat within the submucosal layers of vaginal tissue while keeping the surface cool.

SUMMARY:
This is a prospective, randomized, double-blind, sham-controlled clinical study. The study is designed to demonstrate that active is superior to sham for the efficacy endpoints and is deemed to have appropriate safety as compared to sham.

DETAILED DESCRIPTION:
Approximately ninety-nine (99) subjects meeting the inclusion/exclusion criteria will be randomized in a 2:1 ratio to either the active or sham group. Randomization will be stratified by study site, with a maximum of 21 subjects randomized in an individual site. Subjects will be followed up with at 10 days and at 3 and 6 months post-treatment. Subjects will be assessed for adverse events at all study contacts and visits from the time the informed consent is signed.

ELIGIBILITY:
Key Inclusion Criteria:

* Signed and dated ICF
* Pre-menopausal females
* Documented diagnosis of SUI

Exclusion Criteria:

* Pregnant or planning to become pregnant within the year
* Undergone other SUI treatments (excluding Kegels)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2019-07-05 (Actual); Study Completion 2019-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stacie Bell, PhD, Study Director — Viveve Inc.
Locations (6):
- Canada (6):
  - LIBERATE In't Site, Vancouver, British Columbia
  - LIBERATE Int'l Site, Pointe-Claire, Montreal
  - LIBERATE Int'l Site, Burlington, Ontario
  - LIBERATE Int'l Site, London, Ontario
  - LIBERATE Int'l Site, Sarnia, Ontario
  - LIBERATE Int'l Site, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects completed prescreening and screening visits to assess their level of SUI, perform physical exam to assess their condition and collected initial patient reported outcome data.
Groups:
- Active Treatment: Treatment dose
  Viveve Active Treatment: comprised of therapeutic levels of Radiofrequency (90 J/cm2) and Cryogen Cooling (35 ms pulse).
- Sham Treatment: Sub-therapeutic dose
  Viveve Sham Treatment: comprised of non-therapeutic level of Radiofrequency (<1 J/cm2) and Cryogen Cooling (35 ms pulse).
Period: Overall Study
Arm/Group | Active Treatment | Sham Treatment
Started | 66 (First subject enrolled 8/8/2018. Last subject, last visit, 7/5/2019) | 33 (First subject enrolled 8/8/2018. Last subject, last visit, 7/5/2019)
Completed | 57 | 29
Not Completed | 9 | 4
Not completed — Lost to Follow-up | 3 | 0
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Pregnancy | 1 | 1
Not completed — Discomfort during treatment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active: Viveve Active Treatment: comprised of therapeutic levels of Radiofrequency (90 J/cm2) and Cryogen Cooling (35 ms pulse).
- Sham: Viveve Sham Treatment: comprised of non-therapeutic level of Radiofrequency (<1 J/cm2) and Cryogen Cooling (35 ms pulse).
- Total: Total of all reporting groups
Arm/Group | Active | Sham | Total
Number analyzed (Participants) | 66 | 33 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] — Age in years, including full years and tenths of years was collected
  years | 42.8 (5.51) | 42.3 (4.67) | 42.6 (5.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 33 | 99
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  White | 59 | 30 | 89
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  Canada | 66 | 33 | 99
1 Hour Pad Weight [Median (Inter-Quartile Range); unit: grams] — The 1-hour Pad Weight Test was published by Khrut in 2014). It is a 60 minute procedure that measures the severity of urinary incontinence. It consists of the following:
  1. Subject puts on one standardized, pre-weighed pad without voiding.
  2. Subject drinks 500 mL of water while sitting or resting.
  3. Subject walks for 30 minutes, including climbing one flight of stairs.
  4. Standing up from sitting
  5. Coughing vigorously
  6. Running on the spot 7 Bending to pick up an object from the floor
  The weight of the pad is measured to determine the amount of leakage.
  grams | 12.8 [7.4 to 25.2] | 12.9 [7.6 to 20.4] | 12.9 [7.6 to 23.5]
Urinary Distress Inventory (UDI6) [Median (Inter-Quartile Range); unit: units on a scale] — UDI-6 contains 6 items about urinary problems. Each item is scored between 0 (no problem) to 3 (bothered greatly). All scores are summed, divided by 18 and then multiplied by 100 for the scale score. Minimum scale score is 0 and maximum is 100. Higher scores indicate higher disability.
  units on a scale | 55.6 [44.4 to 66.7] | 55.6 [44.4 to 66.7] | 55.6 [44.4 to 66.7]

OUTCOME MEASURES:

1. Primary Outcome: CFB in 1-hour Pad Weight Test
Description: Change from baseline in the 1-hour pad weight test to 6 months post-treatment.
Time Frame: 6 months post-treatment
Population: Full Analysis Set: randomized subjects in the with non-missing values at the timepoint.
Measure: Median (Inter-Quartile Range); unit: grams
Arm/Group | Active | Sham
Number analyzed (Participants) | 56 | 29
grams | -8.1 [-18.5 to -5.7] | -8.1 [-16.6 to -4.4]

2. Secondary Outcome: Safety and Adverse Event Reporting
Description: Safety as assessed by Adverse Event reporting
Time Frame: 6 months post-treatment
Population: Adverse events are reported in the AE section.
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Sham
Number analyzed (Participants) | 66 | 33
Participants | 24 | 14

3. Other Pre Specified Outcome: UDI-6
Description: Validated urinary incontinence questionnaire titled Urogenital Distress Inventory-6 (UDI-6). UDI-6 contains 6 items about urinary problems. Each item is scored between 0 (no problem) to 3 (bothered greatly). All scores are summed, divided by 18 and then multiplied by 100 for the scale score. Minimum scale score is 0 and maximum is 100. Higher score indicates higher disability. Efficacy measure of change from baseline to 3- and 6- months post-treatment in UDI-6.
Time Frame: 6 months post-treatment
Population: Full Analysis Set: randomized subjects non-missing values at the timepoint.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Active | Sham
Number analyzed (Participants) | 56 | 29
units on a scale | -22.2 [-38.9 to -5.6] | -16.7 [-33.3 to -5.6]

4. Other Pre Specified Outcome: ICIQ-UI-SF
Description: Validated urinary incontinence questionnaire titled International Consultation on Incontinence Modular Questionnaire-Urinary Incontinence Short Form (ICIQ-UI-SF)
Time Frame: 6 months post-treatment
Reporting Status: Not Posted

5. Other Pre Specified Outcome: I-QOL
Description: Validated urinary incontinence questionnaire titled Incontinence Quality of Life (I-QOL)
Time Frame: 6 months post-treatment
Reporting Status: Not Posted

6. Other Pre Specified Outcome: FSFI
Description: Validated questionnaire titled The Female Sexual Function Index (FSFI)
Time Frame: 6 months post-treatment
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Voiding Episodes Per Day
Description: Voiding episodes per day tracked via daily voiding diary.
Time Frame: 6 months post-treatment
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Treatment Emergent Adverse Events reporting occurred from the treatment procedure to study completion (up to 6 months post treatment) for each subject.
Description: Treatment emergent adverse events were evaluated in 66 Active Treatment subjects and 33 Sham Treatment subjects.
Arm/Group | Active Treatment | Sham Treatment
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/33
Serious Adverse Events (participants affected / at risk) | 2/66 | 1/33
Other Adverse Events (participants affected / at risk) | 0/66 | 2/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Treatment (N=66) | Sham Treatment (N=33)
Right Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Subject received active treatment. Experienced a right ankle fracture 50 days after treatment that resulted in hospitalization. The event was coded as unrelated.
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0) — Subject received active treatment. Experienced Angina Pectoris 108 days after treatment which resulted in hospitalization. Event coded as not related.
Freeman-Sheldon Syndrome (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) — Subject was treated with Sham. Became pregnant during the trial and delivered a child with Freeman-Sheldon Syndrome. Pregnancy occurred approximately 60 days post treatment and was coded as not related.
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Treatment (N=66) | Sham Treatment (N=33)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (33)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-10-23): https://cdn.clinicaltrials.gov/large-docs/74/NCT03619174/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-03): https://cdn.clinicaltrials.gov/large-docs/74/NCT03619174/SAP_001.pdf
  • Informed Consent Form (2018-10-31): https://cdn.clinicaltrials.gov/large-docs/74/NCT03619174/ICF_003.pdf